CLINICAL TRIAL: NCT06960265
Title: A Pilot Study for the Effects of Repetitive Transcranial Magnetic Stimulation in Patients With Amphetamine Use Disorders: Clinical Outcomes, Near InfraRed Spectroscopy, and Biomarkers
Brief Title: Effects of Repetitive Transcranial Magnetic Stimulations in Patients With Amphetamine Use Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TsaoTun Psychiatric Center, Department of Health, Taiwan (Other)
Responsible Party: Principal Investigator, Ching-Hua Julie Lee, Attending Psychiatrist, TsaoTun Psychiatric Center, Department of Health, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11457
Record Dates: First submitted 2025-04-20; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Amphetamine Use Disorders; Amphetamine Use Disorder; Amphetamine Dependence; Amphetamine Abuse; NIRS; rTMS; rTMS Stimulation
Keywords: amphetamine; rtms; NIRS
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Controlled (Sham Comparator): The sham group will undergo a placebo procedure using the same rTMS parameters but with a figure-of-eight sham coil, following precedents set by studies on cocaine use disorder treatment (Terraneo et al., 2016).
  Interventions: Device: sham for repetitive Transcranial Magnetic Stimulation
- rTMS treatment group (Experimental): rTMS will be administered at a frequency of 15Hz, with each pulse at 100% rMT intensity. Sessions include 60 pulses per train, with a 26-second inter-train pause, across 40 trains, totaling 2400 pulses over a 20-minute session. Schedule: Participants will receive daily rTMS sessions for the first five days, followed by 5 more sessions for the second week, totaling 10 sessions
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation (rTMS) — Targeting: The left dorsolateral prefrontal cortex (DLPFC) will be the target for treatment.
  Equipment: rTMS will be delivered using a Magstim super rapid magnetic stimulator with a 70-mm air-cooled figure-eight-shaped coil. Resting Motor Threshold (rMT) Measurement: rMT is determined through visual twitch responses in the contralateral hand, identifying the minimal intensity needed to elicit thumb movement in 50% of trials.
  rTMS will be administered at a frequency of 15Hz, with each pulse at 100% rMT intensity. Sessions include 60 pulses per train, with a 26-second inter-train pause, across 40 trains, totaling 2400 pulses over a 20-minute session.
  Arms: rTMS treatment group
Device: sham for repetitive Transcranial Magnetic Stimulation — The sham group will undergo a placebo procedure using the same rTMS parameters but with a figure-of-eight sham coil, following precedents set by studies on cocaine use disorder treatment (Terraneo et al., 2016).
  Arms: Controlled

SUMMARY:
Amphetamine Use Disorder (AUD) is a major public health issue in Taiwan, where it is the most commonly abused illegal drug. There are currently no effective approved medications to treat it, which makes finding new treatment options urgent. Repetitive Transcranial Magnetic Stimulation (rTMS), a non-invasive brain stimulation method, has shown promise in reducing cravings and drug use in people with addiction, but its effects on AUD are not well studied.

To explore this, the investigators plan to conduct a double-blind, sham-controlled study with 20 people diagnosed with AUD. Half will receive real rTMS treatment, and half will receive a placebo-like sham treatment. The treatment targets a specific brain area (the left dorsolateral prefrontal cortex) and will be given 10 times over two weeks.

The investigators will assess the effectiveness of rTMS by tracking drug cravings, urine test results, and side effects with follow-up over 12 weeks. The investigators also include brain imaging using near-infrared spectroscopy (NIRS) after the treatment.

The study aims to better understand how rTMS might help reduce amphetamine cravings and improve outcomes, potentially leading to new treatment options for AUD.

DETAILED DESCRIPTION:
Amphetamine Use Disorder (AUD) is a serious and growing public health concern, especially in Taiwan, where amphetamines are the most commonly misused illegal drugs. Globally, amphetamines also rank among the top drugs of abuse. Despite the widespread impact of this condition, there are currently no approved medications that effectively treat amphetamine addiction. This gap in treatment options underscores the urgent need for new and innovative approaches to help individuals struggling with AUD.

One promising method being explored is Repetitive Transcranial Magnetic Stimulation (rTMS). This is a non-invasive technique that uses magnetic fields to stimulate specific areas of the brain. It has already shown positive effects in treating several mental health conditions, such as depression and anxiety, and early studies suggest it may also help reduce cravings and drug use in people with substance use disorders.

This study aims to investigate whether rTMS can help people with AUD by reducing their cravings and improving their chances of recovery. To do this, the investigators will conduct a carefully controlled clinical trial involving 20 participants who have been diagnosed with AUD. The participants will be randomly divided into two groups. One group will receive active rTMS treatment, while the other will receive a "sham" or placebo version of the treatment. This means the second group will undergo the same procedure without the magnetic stimulation, allowing us to accurately measure the true effects of rTMS.

The treatment will focus on a brain area called the left dorsolateral prefrontal cortex (DLPFC), which is involved in decision-making, impulse control, and craving regulation. The rTMS sessions will use a high-frequency setting (15 Hz) delivered in short bursts, with a total of 10 sessions spread over two weeks.

To understand the impact of the treatment, the investigators will collect several types of data from participants throughout the study (pre and post) and for 12 weeks afterward. This includes:

Urine drug tests to check for ongoing amphetamine use Craving assessments to see if the urge to use drugs decreases Monitoring for side effects to ensure safety Neuropsychological tests to assess changes in thinking and behavior Brain imaging using near-infrared spectroscopy (NIRS) to observe changes in brain activity Through this comprehensive approach, the investigators hope to learn more about how rTMS works in the context of amphetamine addiction and whether it could be developed into an effective treatment. The findings could pave the way for new, science-based therapies to support individuals with AUD and reduce the burden of this condition on individuals, families, and society.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years.
* Meeting DSM-5 criteria for substance use disorder made by a specialist in addiction psychiatry.
* Fluency in Chinese.
* Willingness and ability to comply with study requirements.
* Good physical health determined by complete physical examination, and laboratory tests.
* Patient or a reliable caregiver can be expected to ensure acceptable compliance and visit attendance for the duration of the study.
* Trained psychiatrists will assess eligible patients using the structured clinical interview for the Mini-International Neuropsychiatric Interview (MINI) (Sheehan et al., 1998) to determine the presence of any psychotic disorder.

Exclusion Criteria:

* Evidence of an uncontrolled and/or clinically significant medical condition, e.g., cardiac, hepatic and renal failure that would compromise patient safety or preclude study participation.
* Premorbid mental retardation.
* Other major Axis-I Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) diagnoses other than substance use disorder.
* Pregnancy or nursing.
* History of seizures or epilepsy.
* History of neurological diseases or traumatic brain injury.
* Suicidal attempts or risks during screening or study period.
* Presence of prosthesis devices, e.g. pace-makers, cochlear prosthesis, neuro- stimulators, magnetic cochlear prosthesis, intraocular metallic fragments.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Average Hb level using Near-infrared spectroscopy (NIRS) | From enrollment to the end of treatment at 2 weeks.
  NIRS will focus on oxy-Hb and deoxy-Hb of frontal lobe and left and right sides frontal lobe. Later the average Hb will be calculated for frontal lobe and left and right sides frontal lobe.
Urine Drug Test | From enrollment to the end of treatment at 2 weeks and at 3 months follow up.
  Urine drug tests to check for ongoing amphetamine use

SECONDARY OUTCOMES:
Amphetamine Dependence Level | From enrollment to the end of treatment at 2 weeks and at 3 months follow up.
  Severity of Dependence Scale (SDS) (V. C. H. Chen et al., 2008)
Amphetamine Craving Level | From enrollment to the end of treatment at 2 weeks and at 3 months follow up.
  Craving Scale: Includes the Drug-Use and Craving Questionnaire (Huang et al., 2021)
Impulsivity Level | From enrollment to the end of treatment at 2 weeks and at 3 months follow up.
  Barratt Impulsiveness Scale (BIS-11) (Patton et al., 1995)
Level for Quality of Life | From enrollment to the end of treatment at 2 weeks and at 3 months follow up.
  WHO Quality of Life instrument - BREF (WHOQOL-BREF) (Yao et al., 2002)
Anxiety Level | From enrollment to the end of treatment at 2 weeks and at 3 months follow up.
  General Anxiety Disorder-7 (GAD-7) (Spitzer et al., 2006)
Depression Level | From enrollment to the end of treatment at 2 weeks and at 3 months follow up.
  Chinese Version of the Centre for Epidemiologic Studies Depression Scale (CESD- C) (Cheng & Chan, 2005; Radloff, 1977)
Erectile Function | From enrollment to the end of treatment at 2 weeks and at 3 months follow up.
  International Index of Erectile Function (IIEF-5) (Rosen et al., 1998)
Suicidality | From enrollment to the end of treatment at 2 weeks and at 3 months follow up.
  Ask Suicide-Screening Questions (ASQ) (Horowitz et al., 2012)

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hua Julie Lee, MD., MPH, Principal Investigator — Tsaotun Psychiatric Center, Ministry of Health and Welfare
Locations (1):
- TsaoTun Psychiatric Center, Nantou City, Taiwan

IPD SHARING:
Plan to Share IPD: No